CLINICAL TRIAL: NCT06394583
Title: DESCRIPTION OF THE LUNG ULTRASOUND PATTERN IN INFANTS UNDER 26 WEEKS OF GESTATION: A NATIONAL MULTICENTER STUDY
Brief Title: LUS AT BIRTH IN INFANTS BORN BEFORE 26 WEEKS
Acronym: MINI-LUS
Status: Not yet recruiting | Type: Observational
Sponsor: Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, Almudena Alonso Ojembarrena, MD, PhD, Andaluz Health Service
Other Study IDs: NEO-LUS-24-01
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Extremely Low Birth Weight Infants; Respiratory Distress Syndrome, Newborn
Keywords: lung ultrasound; premature infant; extremely low birth weight infants
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Lung ultrasound — We will perform a LU at birth to all infants, before the first dose of surfactant.

SUMMARY:
All infants born before 26 weeks born in a hospital included in the registry will receive a LU at birth, before the first dose of surfactant. We will register as well the length of IMV, NIV or the need of IMV in the whole sample.

ELIGIBILITY:
Inclusion Criteria:

* Infants born before 26 weeks at any of the participant hospitals.

Exclusion Criteria:

* received surfactant before LU
* redirection of care
* severe malformations of cromosomopathies
* unable to perform LU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants born before 26 weeks in any of the centers included in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Description of LU patterns | at birth

SECONDARY OUTCOMES:
need of IMV | during NICU admission
length of IMV | during NICU admission
length of NIV | during NICU admission

IPD SHARING:
Plan to Share IPD: No
Each investigator will review only the data from their own hospital.